CLINICAL TRIAL: NCT06554964
Title: Feasibility, Safety and Effectiveness of Chromotubation on the Remaining Fallopian Tube After a Laparoscopic Salpingectomy Due to Tubal Pregnancy
Brief Title: Chromotubation on the Remaining Fallopian Tube After a Laparoscopic Salpingectomy Due to Tubal Pregnancy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Neta Eisenberg Kogan, Attending physician in the gynecology endoscopy unit, Assaf-Harofeh Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0135-24-ASF
Record Dates: First submitted 2024-08-08; First posted 2024-08-15 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Intervention Model Description: Prospective non-randomized cohort study including patients undergoing laparoscopic salpingectomy for tubal ectopic pregnancy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing laparoscopic salpingectomy for tubal ectopic pregnancy. (Experimental): Patient undergoing laparoscopic salpingectomy due to ectopic tubal pregnancy will be offered chromotubation as the same tome in order to asess the potency of the remaining fallopian tube. Data will be recorded.
  Interventions: Procedure: performing chromotubation during the laparoscopy in order to assess the tubal patency of the remaining fallopian tube

INTERVENTIONS:
Procedure: performing chromotubation during the laparoscopy in order to assess the tubal patency of the remaining fallopian tube — Performing chromotubation )injection of blue dye to the fallopian tube via cevical catheter) during the laparoscopy in order to assess the tubal patency of the remaining fallopian tube

SUMMARY:
Ectopic pregnancy prevalence is approximately 1-2% of all pregnancies, majority of which located in the fallopian tube. Among the risk factors for ectopic pregnancy is tubal factor - meaning a mechanical problem within the fallopian tube resulting in the pregnancy remaining in the fallopian tube. The treatment o tubal pregnancy can be expectant, medical via metotrexate or surgicl via laparoscopic salpingectomy of the involved fallopian tube. The purpose of this study is to assess the feasibility of chromotubation during laparoscopic salpingectomy for the surgical management of tubal ectopic pregnancy hence assessing the function of the remaining fallopian tube and trying to predict future fertility for the patient.

DETAILED DESCRIPTION:
Ectopic pregnancy occurs approximately in 1-2% of all pregnancies. The risk is higher among patients with risk factors such as previous ectopic pregnancy, history of pelvic inflammatory disease, endometriosis, past tubal surgery, pregnancy following in vitro fertilization, and pregnancy conceived with an intrauterine device. In 97% of the cases the location of the ectopic pregnancy would be in the fallopian tube. The management of fallopian tube ectopic pregnancy can be expectant, medical (with intramuscular methotrexate) or surgical via laparoscopic salpingectomy of the involved fallopian tube. The optimal management is chosen depending on the clinical presentation, sonographic and laboratory findings and patient's wishes.

Laparoscopic salpingectomy is indicated in cases of suspected ruptured ectopic pregnancy. Salpingectomy is also offered in cases of recurrent ipsilateral ectopic pregnancy, contraindications to medical management with methotrexate, and patients who prefer surgical over medical treatment.

The risk of recurrent ectopic tubal pregnancy following unilateral laparoscopic salpingectomy varies according to the functionality of the remaining fallopian tube and between different studies. In cases of an abnormal contralateral fallopian tube, the risk of recurrent tubal pregnancy is high. For patients with a healthy contralateral fallopian tube some studies found that the long-term fertility after salpingectomy was not significantly impacted, while other studies reported a mild reduction in natural conception rates. Thus, it is estimated that a functional remaining fallopian tube may capture oocytes from both ovaries, and may compensate for the loss of the other fallopian tube. Overall, the patency and functionality of the remaining fallopian tube is the most important factor in determining the risk of recurrent ectopic pregnancy and the rates of subsequent natural intrauterine conception.

Chromotubation is a procedure used in order to assess the patency of the fallopian tubes, mostly at time of laparoscopy under general anesthesia. It involves the injection of colored blue dye (mostly methylene blue or indigo carmine) through the cervix and into the uterine cavity and the fallopian tubes. During laparoscopy, the flow of the dye through the fallopian tubes may be observed, and the patency of the fallopian tubes may be determined.

The intracervical use of methylene blue or indigo-carmine for laparoscopic chromotubation is generally considered safe. Rare adverse reactions were described among patients with G6PD deficiency for whom methylene blue may cause hemolysis and for patient who are treated with SSRI for whom methylene blue may cause serotonin toxicity due to inhibition of monoamine oxidase.

Other methods to evaluate the patency of the fallopian tubes include hysterosalpingogram (HSG) and ultrasound guided perturbation using Exfoam. These imaging procedures are performed without anesthesia (and may be associated with pain and discomfort), and their results may be inconclusive because of tubal spasm. Thus laparoscopic chromotubation, which allows for the evaluation of tubal patency and pelvic anatomy, is considered the gold standard procedure.

The current practice in the management of patients undergoing laparoscopic salpingectomy for tubal pregnancy includes observation of the pelvic and tubal anatomy at time of surgery, followed by referral for outpatient assessment of tubal patency by HSG or by ultrasound at a later date, usually after ~2 months.

In the current study, the investigators propose to perform an evaluation of tubal patency by laparoscopic chromotubation at time of laparoscopic salpingectomy for tubal pregnancy. The investigators will assess the feasibility of the procedure (i.e., whether tubal patency may be determined in this setting), and its safety.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing laparoscopic salpingectomy for tubal ectopic pregnancy.

Exclusion Criteria:

1. Patients with a history of unilateral salpingectomy
2. Patients with suspected heterotopic pregnancy
3. Patients with suspected allergic reaction to blue dye injection

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The subjects in this study are patients with ectopic pregnancy hence are females
Enrollment: 100 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Precentage of successful chromotubation (passing of blue dye through the fallopian tube) during laparoscopic salpingectomy for the surgical management of tubal ectopic pregnancy. | 1 year
  How many cases would demonstrate patent fallopian tube via blue dye injected verses how many occluded ones.

SECONDARY OUTCOMES:
Percentage of adverse reaction to chromotubation during laparoscopic salpingectomy for the surgical management of tubal ectopic pregnancy. | 1 year
  How many allergic reactions

CONTACTS AND LOCATIONS:
Overall Officials: Neta Eisenberg-Kogan, MD, Principal Investigator — Assaf-Harofeh Medical Center

IPD SHARING:
Plan to Share IPD: Yes
date will be shared and published once study is complected
Supporting Information: CSR
Time Frame: date will be shared once study is complected for unlimited time
Access Criteria: date will be shared in relevant publications